CLINICAL TRIAL: NCT02972853
Title: Mindfulness Influences on Self-Regulation: Mental and Physical Health Implications: Mindful Self-Regulation fMRI Pilot Study
Brief Title: Mindful Self-Regulation fMRI Pilot Study
Acronym: MindfulPCMRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cambridge Health Alliance (Other)
Collaborators: Martinos Center for Biomedical Imaging (Other); National Center for Complementary and Integrative Health (NCCIH) (NIH); Brown University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CHA-IRB-1002/08/14; 1UH2AT009145-01 (NIH)
Record Dates: First submitted 2016-11-16; First posted 2016-11-25 (Estimated); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Psychiatric Problem; Depression; Anxiety; Neuroimaging; Self-Control
MeSH Terms: conditions — Depression; Anxiety Disorders; Self-Control | interventions — Primary Health Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mindfulness Training for Primary Care (Experimental): For intervention description see Mindfulness Training for Primary Care (MTPC) in the study "MINDFUL-PC: Integrating Mindfulness Into the Patient-Centered Medical Home - A Pilot Study". For the Mindfulness Training for Primary Care (MTPC) fMRI - arm, we acquire pre-/post-intervention neuroimaging measures from subjects enrolled in this additional pilot fMRI study.
  Interventions: Behavioral: Mindfulness Training for Primary Care (MTPC)

INTERVENTIONS:
Behavioral: Mindfulness Training for Primary Care (MTPC) — For intervention description see Mindfulness Training for Primary Care (MTPC) in the study "MINDFUL-PC: Integrating Mindfulness Into the Patient-Centered Medical Home - A Pilot Study"

SUMMARY:
The purpose of this study is to 1) determine whether Mindfulness Training for Primary Care (see study "MINDFUL-PC: Integrating Mindfulness Into the Patient-Centered Medical Home - A Pilot Study") engages self-regulation targets such as emotion regulation, attention, and interoceptive awareness; and 2) changes brain activation in neuroimaging tasks before compared to after the training. Neuroimaging fMRI tasks probe mechanisms related to self-regulation, such as attention/inhibition, emotion regulation, self-compassion, interoception and pain regulation.

The study will also look at whether chronic disease self-management and successful engagement of self-report and behavioral self-regulation targets (emotion regulation, attention, and interoceptive awareness) relates to the observed brain activation changes after compared to before the mindfulness intervention.

DETAILED DESCRIPTION:
This study aims to test brain activation changes related to self-regulation targets of attention, emotion regulation, self-compassion, interoception and pain regulation that are influenced by mindfulness training within primary care (compare MINDFUL-PC study).

The study will also look at whether successful chronic disease self-management relates to the observed brain activation changes after compared to before the mindfulness intervention.

The study will examine the relationship between mindfulness training within primary care and medical regimen adherence (initiation and maintenance) as well as the underlying neural correlates associated with changes in self-regulation.

This is a single-arm pilot trial, recruiting from a randomized controlled trial (see MINDFUL-PC study). .

ELIGIBILITY:
Inclusion Criteria:

* Adults 21-60 years old enrolled for participation in the MINDFUL-PC study.
* During baseline visit, patient has a history of either major depressive disorder, dysthymia, or generalized anxiety disorder, OR has current mild to moderate symptoms of depression (score range of 10-28 on DASS-21 Depression subscale) or anxiety (score >7 on DASS-21 anxiety subscale).
* Participant does not have a substance use disorder nor intoxication at the time of scanning. Participants must report no more than infrequent recreational cannabis use (i.e., no more than two times a month) and must report capacity for abstinence from both cannabis and ethyl alcohol for the 72 hours prior to the scan.
* Normal or corrected-to-normal vision, and correction must be with contact lenses.
* Right-handed as defined by Edinburgh Handedness Inventory.

Exclusion Criteria:

* Current severe panic disorder, active severe PTSD symptoms, or psychosis.
* Current suicidality OR severe depression as evidenced by a score of 28 or higher on the DASS-21 Depression subscale.
* Standard direct exclusion criteria for undergoing magnetic resonance imaging (MRI) procedures for research purposes (safety standards), i.e., Meniere's disease, epilepsy, strong claustrophobia, currently pregnant or breastfeeding or planning to conceive or breastfeed during the study, cardiac pacemaker, prosthetic heart valve, neurostimulator, implanted pumps, non-MR-compatible implants or devices.
* A history of neurological disease or injury, including a history of seizures or significant head trauma (i.e., extended loss of consciousness, neurological sequelae, or known structural brain lesion), or previous brain surgery.
* Severe skin disease, skin allergies, or multiple reactions to topical preparations, dressings or tapes.
* Current meditation or intense yoga practice or extensive previous experience.
* Participants with vascular disease, such as peripheral vascular disease, varicose veins, or lymphedema, in both lower limbs.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2020-10 (Actual)

PRIMARY OUTCOMES:
Change in Brain activation in regions of interest | 8 weeks
  Change in brain activation will be measured with functional magnetic resonance imaging (fMRI) during four different tasks: an affective go/nogo regulation task, an interoceptive attention task, a self-compassion task and a pain regulation task. Brain activation will be compared between baseline and Week 8.

SECONDARY OUTCOMES:
Correlations between brain activation changes and self-regulation measures | 8 weeks
  Self-regulation targets of emotion regulation, interoceptive awareness, and attention from MINDFUL-PC: Integrating Mindfulness Into the Patient-Centered Medical Home."
Correlations between brain activation changes and chronic disease self-management action plan initiation. | 9 weeks
  In addition, brain activation in regions of interest will be correlated with chronic disease self-management action plan initiation.

CONTACTS AND LOCATIONS:
Overall Officials: Zev D Schuman-Olivier, MD, Principal Investigator — Cambridge Health Alliance
Locations (1):
- CHA Center for Mindfulness and Compassion, Somerville, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No